CLINICAL TRIAL: NCT04302220
Title: Natural History of Myopic Optic Neuropathy for High Myopia in Chinese Adult Population: a Registry Cohort Study
Brief Title: Myopic Optic Neuropathy in Chinese High Myopia Population
Status: Active, not recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiulan Zhang, Professor of Ophthalmology, Director of Clinical Research Center, Director of CFDA-certified Pharmaceutical Research Unit, State Key Laboratory of Ophthalmology, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2019KYPJ079
Record Dates: First submitted 2020-03-07; First posted 2020-03-10 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Eye Diseases
Keywords: myopic optic neuropathy; high myopia; glaucoma
MeSH Terms: conditions — Eye Diseases; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Saliva smple.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- high myopia: Population who have high myopia.

SUMMARY:
This study intends to establish a registry cohort to enroll patients with high myopia to study the natural course of myopic optic neuropathy in Chinese adult population.

DETAILED DESCRIPTION:
Global prevalence of high myopia brings about markedly increasing of blinding complications as myopic optic neuropathy (MON) and glaucoma. It was estimated that there were 163 million people who have high myopia in 2000, and the population with high myopia would increase to almost one billion (9.8% of the world population) worldwide by 2050.

Glaucoma is the leading cause of irreversible blindness worldwide while it is difficult to distinguish glaucoma among MON in high myopia eyes. However, there lack longitudinal study to illustrate the natural course interpreting the distribution and natural history of MON.

In view of the above problems, this is a longitudinal registry cohort study to observe the long-term changes of structural and functional parameters of MON in high myopia, and to investigate the natural course and associted risk factors that influence the progression in a Chinese adult population.

ELIGIBILITY:
Inclusion Criteria

* Age ≥18 years
* Equivalent spherical ≤-6D or axial length ≥26.5mm
* Best corrected visual acuity ≥ 6/12

Exclusion Criteria

* Unwilling or unable to give consent, or unable to return for scheduled protocol visits.
* Glaucoma secondary to penetrating keratoplasty, trauma, steroids, retinal disease/surgery, or neovascular disease.
* Obvious corneal and iris lesions, or severe cataracts interfering with fundus examinations, VF test or monophthalmia.
* Need for ocular surgery/laser or anticipated need for cataract surgery during the study period.
* Other serious systemic diseasesf (i.e. hypertension, heart disease, diabetes, or rheumatic immune system diseases);
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have high myopia aged from 18 to above.
Sampling Method: Non-Probability Sample
Enrollment: 813 (Estimated)
Dates: Start 2019-06-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression of glaucoma within 36 months | 3 years
  Structural and functional changes of glaucoma using visual field, stereoscopic fundus photography.

SECONDARY OUTCOMES:
Progression of myopia and other structural changes of retina and choroid. | 3 years
  Structural and functional changes of myopia based on axial length and refractive error.

CONTACTS AND LOCATIONS:
Overall Officials: Xiulan Zhang, MD, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Lin F, Chen S, Song Y, Li F, Wang W, Zhao Z, Gao X, Wang P, Jin L, Liu Y, Chen M, Liang X, Yang B, Ning G, Cheng CY, Healey PR, Park KH, Zangwill LM, Aung T, Ohno-Matsui K, Jonas JB, Weinreb RN, Zhang X; Glaucoma Suspects with High Myopia Study Group. Classification of Visual Field Abnormalities in Highly Myopic Eyes without Pathologic Change. Ophthalmology. 2022 Jul;129(7):803-812. doi: 10.1016/j.ophtha.2022.03.001. Epub 2022 Mar 12. PMID 35288144
- [Derived] Song Y, Wang W, Lin F, Chen S, Jin L, Li F, Gao K, Cheng W, Xiong J, Zhou R, Chen M, Liang J, Zhang J, Jonas JB, Zhang X. Natural history of glaucomatous optic neuropathy in highly myopic Chinese: study protocol for a registry cohort study. BMJ Open. 2020 Dec 30;10(12):e039183. doi: 10.1136/bmjopen-2020-039183. PMID 33380478